CLINICAL TRIAL: NCT00892853
Title: Association of Bone Quality and Quantity With Vascular Calcification.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yebin Jiang, M.D., Primary Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 00022370
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Vascular Calcification; Atherosclerosis; Bone Density
Keywords: calcification; osteoporosis
MeSH Terms: conditions — Vascular Calcification; Atherosclerosis; Calcinosis; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone Density Scanning (Other): To acquire high resolution images of the bones and aid in determining bone density.
  Interventions: Procedure: CT of the bones

INTERVENTIONS:
Procedure: CT of the bones — A CT scan will be performed on one arm and one leg for the purpose of acquiring images for this research study.

SUMMARY:
The purpose of this study is to determine if there is a link between calcium build up in the veins or arteries (including the veins/arteries of the heart) and deterioration of the bone. This will help understand if there is a connection between heart disease and bone disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 30 years of age or older
* Must already be scheduled to have a CT examination of the arteries of the heart

Exclusion Criteria:

* Diagnosed with bone cancer
* Previous diagnosis of cancer that's spread to the bone
* History of cancer that involves bone marrow
* Any bone disease other than osteoporosis
* Any disease which leads to serious osteoporosis or vascular calcification such as:

  * kidney disease
  * thyroid and adrenal disease
  * anorexia nervosa
  * secondary osteoporosis

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To determine if there is a connection between heart disease and bone disease through correlation of bone density with the calcium deposited in the coronary arteries. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yebin Jiang, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States